CLINICAL TRIAL: NCT02191527
Title: Evaluating the Effectiveness of Point-of-care Diagnostic Technologies in MCH Services and Their Impact on Mother and Child Health Outcomes in Cabo Delgado Province, Mozambique
Brief Title: Evaluating the Effectiveness of Point-of-care Diagnostic Technologies in MCH Services in Mozambique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Ministry of Health, Mozambique (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EGPAF-004
Record Dates: First submitted 2013-08-15; First posted 2014-07-16 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: HIV; Syphilis; Anemia During Pregnancy
Keywords: PMTCT; HIV; Syphilis; Anemia during pregnancy; Point of care diagnostics
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Intervention Model Description: Before and after intervention study design
Oversight: Data Monitoring Committee: No

ARMS (2):
- Point of Care Testing (Experimental): The point-of-care devices will be located in the MCH services, where a trained lay counselor will do the tests.
  Interventions: Device: PIMA® for quantitative analysis of CD4-count; Device: Hemocue® (HemoCue AB, Angelhom, Sweden) for quantitative analysis of hemoglobin; Device: SD Bioline® (Standard Diagnostics Inc., South-Korea) for qualitative analysis of syphilis
- Laboratory Testing - Standard of care (No Intervention): Samples sent to the laboratory for analysis, (standard of care)

INTERVENTIONS:
Device: PIMA® for quantitative analysis of CD4-count
  Arms: Point of Care Testing
Device: Hemocue® (HemoCue AB, Angelhom, Sweden) for quantitative analysis of hemoglobin
  Arms: Point of Care Testing
Device: SD Bioline® (Standard Diagnostics Inc., South-Korea) for qualitative analysis of syphilis
  Arms: Point of Care Testing

SUMMARY:
The general goal of the proposed study is to evaluate the cost-effectiveness of POC technologies for diagnosis of syphilis, quantitative analysis for hemoglobin and CD4 counting performed within MCH services to improve maternal and infant health.

A prospective, quasi-experimental study will be done in Cabo Delgado province, where health facilities will be randomized in an intervention or comparison arm. Outcomes on maternal and infant health will be measured.

ELIGIBILITY:
Inclusion Criteria:

* First antenatal care visit
* Able to provide informed consent and signed consent form
* Minimum 18 years of age
* Diagnosed HIV positive at antenatal care visit
* Living in the catchment area of the health facility

Exclusion Criteria:

* Age <18 years
* No consent form signed
* Being on ART at time of first antenatal care visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1673 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The proportion of HIV positive pregnant women initiating antiretroviral therapy among eligible women. | Within 1 month
  Number of HIV positive pregnant women initiating antiretroviral therapy divided by the number of eligible HIV positive pregnant women

SECONDARY OUTCOMES:
Proportion of women at first ANC visit tested and treated for syphilis | Within 1 month
  Number of women at first ANC tested and treated for syphilis divided by the number of women attending first ANC visit
The proportion of pregnant women tested and treated for anemia | Within 1 month
  Number of pregnant women test and treated for anemia divided by the number of pregnant women
Number of HIV infections in infants averted | 1-3 months of age
  Number of HIV-positive pregnant women who accessed antiretrovial therapy in a timely manner

CONTACTS AND LOCATIONS:
Overall Officials: Caroline DeSchacht, MD, MSc, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation; Ilesh V Jani, MD, PhD, Principal Investigator — Instituto Nacional de Saúde, Mozambique